CLINICAL TRIAL: NCT04751045
Title: Comparison and Outcomes of Endoscopic Ultrasound Liver Biopsies Versus Percutaneous Liver Biopsies: A Randomized Clinical Trial
Brief Title: Comparison and Outcomes of Endoscopic Ultrasound Liver Biopsies Versus Percutaneous Liver Biopsies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Ghassan M. Hammoud, Professor of Clinical Medicine, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013389
Record Dates: First submitted 2020-12-02; First posted 2021-02-11 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Intervention Model Description: Study the safety, efficacy of EUS guided liver biopsy in comparison to percutaneous liver biopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Liver biopsy (Active Comparator): Technique: The preprocedure "time out" protocol will be completed prior to initiation of the procedure. The patient will be positioned supine and right hepatic lobe was localized with ultrasound. Conscious sedation with Versed and fentanyl will be initiated and the patient's vital signs were monitored by an independent trained observer during the procedure.
  After placing a mark on the skin overlying the right upper quadrant, the skin was then prepped and draped in the usual sterile fashion. Maximum sterile barrier technique used at the procedure. Under direct sonographic guidance, a 15 gauge percutaneous liver biopsy needle will be used with a 2 cm throw was advanced into the right hepatic lobe. The biopsy samples will be obtained and submitted to pathology.
  Interventions: Procedure: EUS liver biopsy
- Endoscopic ultrasound guided liver biopsy (Active Comparator): Procedure details: patients will be screened preoperatively to assess cardiovascular health prior to undergoing procedure as this is standard of care. Patients will follow all standard preoperative instructions prior to anesthesia. Upon undergoing general anesthesia, a videoendoscope will be introduced into the esophagus under direct vision. Once endoscope is in position near the liver, a 19-gauge sharkcore needle will be used to puncture the left lobe with a 3 accentuation and another pass from right lobe with 4 accentuation. Doppler study will be used to interrogate for any significant doppler signals in needle path. Post procedure, patients will be provided instructions to avoid NSAIDs for 4 days and perform lightweight activity for 4 days. Patients will be observed for bleeding and significant abdominal pain postoperatively
  Interventions: Procedure: EUS liver biopsy

INTERVENTIONS:
Procedure: EUS liver biopsy — Endoscopic ultrasound guided liver biopsy

SUMMARY:
Histopathological examination of liver tissue is used to determine the etiology and extent of liver disease. In order for a clinician to make a better-informed decision regarding a patient with liver disease, the liver biopsy specimen has to be adequate and of high quality for pathological interpretation. It is generally agreed that an adequate liver biopsy has to have ≥6-12 intact portal tracts for pathological review and interpretation.(1) Historically, three approaches have been used to obtain a liver biopsy: percutaneous, transjugular (TJ-LB) and laparoscopic approach (LA-LB)- with percutaneous liver biopsy (P-LB) being the most commonly employed. Endoscopic ultrasound-guided liver biopsy (EUS-LB), a newer approach, is now being performed by select skilled endoscopists across the country. EUS-LB is advantageous over existing techniques because it enables visualization and avoidance of vessels that are 1mm in diameter, provides access to both lobes of the liver and theoretically is less painful due to avoiding somatic pain fibers. Further, in patients that are already undergoing esophagogastroduodenoscopy, EUS-LB can be performed simultaneously and spare the patient an additional procedure. Because of the plausibility of reduced pain, number of procedures and possibly complications, EUS-LB may be cost-effective over existing methods. There is limited data evaluating the safety and efficacy of EUS-LB versus percutaneous liver biopsy.

The investigators hope to provide answers in a prospective study comparing between patients, who are already undergoing liver biopsy, randomly assigned to either EUS-LB or P-LB. The investigators will compare outcomes such as pain, bleeding, hospitalization, and tissue diagnosis between the two groups. This will allow us to add to the existing data for the use of EUS-LB. If patients are found to have less adverse events and better outcomes using EUS-LB versus percutaneous-LB this may become the preferred method of diagnosis in this patient population.

DETAILED DESCRIPTION:
Date: 01/03/2019 Version Number: 1 Principal Investigator: Ghassan Hammoud MD Application Number: 2011629 Application Title: Comparison and Outcomes of Endoscopic Ultrasound Liver Biopsies versus Percutaneous Liver Biopsies: A Randomized Clinical Trial.

Protocol

* Use the section headings to write the Protocol, inserting the appropriate material in each. If a section is not applicable, leave heading in and insert N/A.
* When submitting Protocol (new or revised), enter the date and version number to

Abstract

1. Provide no more than a one-page research abstract briefly stating the problem, the research hypothesis, and the importance of the research.

   Histopathological examination of liver tissue is used to determine the etiology and extent of liver disease. In order for a clinician to make a better-informed decision regarding a patient with liver disease, the liver biopsy specimen has to be adequate and of high quality for pathological interpretation. It is generally agreed that an adequate liver biopsy has to have ≥6-12 intact portal tracts for pathological review and interpretation.(1) Historically, three approaches have been used to obtain a liver biopsy: percutaneous, transjugular (TJ-LB) and laparoscopic approach (LA-LB)- with percutaneous liver biopsy (P-LB) being the most commonly employed. Endoscopic ultrasound-guided liver biopsy (EUS-LB), a newer approach, is now being performed by select skilled endoscopists across the country. EUS-LB is advantageous over existing techniques because it enables visualization and avoidance of vessels that are 1mm in diameter, provides access to both lobes of the liver and theoretically is less painful due to avoiding somatic pain fibers. Further, in patients that are already undergoing EGD, EUS-LB can be performed simultaneously and spare the patient an additional procedure. Because of the plausibility of reduced pain, number of procedures and possibly complications, EUS-LB may be cost-effective over existing methods. There is limited data evaluating the safety and efficacy of EUS-LB versus percutaneous liver biopsy.

   The investigators hope to provide answers in a prospective study comparing between patients, who are already undergoing liver biopsy, randomly assigned to either EUS-LB or P-LB. The investigators will compare outcomes such as pain, bleeding, hospitalization, and tissue diagnosis between the two groups. This will allow us to add to the existing data for the use of EUS-LB. If patients are found to have less adverse events and better outcomes using EUS-LB versus percutaneous-LB this may become the preferred method of diagnosis in this patient population.

   Background (briefly describe pre-clinical and clinical data, current experience with procedures, drug or device, and any other relevant information to justify the research)

   Several studies are emerging on the safety and efficacy of EUS-LB for diagnosis of patients with liver disease, with only one prospective study.(2) Shah et al. published in 2017 after retrospective review that EUS-LB is safe and efficacious in patients for diagnostic evaluation.(3) Diehl et al. evaluated diagnostic yield of EUS-LB and safety finding it to be successful and safe for obtaining adequate biopsies.(2) Nieto's team looked retrospectively at EUS-LB using a specific needle and one pass method finding it to be safe and effective with rare adverse events of abdominal pain and hematoma.(4) Currently, there is a randomized clinical trial at Brigham and Women's Hospital comparing safety and efficacy of EUS-LB vs. P-LB (ClinicalTrials.Gov NCT02947516).

   Our advanced endoscopists, Drs. Hammoud and Samiullah, perform endoscopic ultrasounds regularly for diagnostic and/or therapeutic reasons, as part of the routine standard of care. Doctor Ghassan Hammoud has successfully performed EUS-LB procedures and will be the sole endoscopist performing the EUS-LB for patients in this study. Many patients who are undergoing endoscopic ultrasound exams are referred to the hepatologists at our institution for evaluation of persistently abnormal hepatic enzymes in whom noninvasive workup for liver diseases has failed to unfold the underlying etiology. As a result, liver biopsy for further assessment and evaluation is strongly considered in this subset of patients.

   Study Procedures
2. Study design, including the sequence and timing of study procedures (distinguish research procedures from those that are part of routine care).
3. Study duration and number of study visits required of research participants.
4. Blinding, including justification for blinding or not blinding the trial, if applicable.
5. Justification of why participants will not receive routine care or will have current therapy stopped.
6. Justification for inclusion of a placebo or non-treatment group.
7. Definition of treatment failure or participant removal criteria.
8. Description of what happens to participants receiving therapy when study ends or if a participant's participation in the study ends prematurely.

This is a prospective randomized clinical trial comparing the safety and efficacy of EUS-LB to P-LB. Patients who meet the inclusion criteria will be informed of their options with respect to obtaining the liver biopsy. Patients will be informed of all the risks (perforation, bleeding, infection, adverse effects related to peri-procedural medications, etc.). Those in agreement will provide informed consent to use their de-identified data for diagnosis and research purposes.

This study will run over a year period or up to when the target number of patients are consented whichever comes first. Patients will only be required to visit for the EUS-LB appointment as already scheduled for standard of care. The study will not be blinded to the researchers; however personal identifiers will be removed as data is collected.

Procedure details: patients will be screened preoperatively to assess cardiovascular health prior to undergoing procedure as this is standard of care. Patients will follow all standard preoperative instructions prior to anesthesia. Upon undergoing general anesthesia, a videoendoscope will be introduced into the esophagus under direct vision. Once endoscope is in position near the liver, a 19-gauge sharkcore needle will be used to puncture the left lobe with a 3 accentuation and another pass from right lobe with 4 accentuation. Doppler study will be used to interrogate for any significant doppler signals in needle path. Post procedure, patients will be provided instructions to avoid NSAIDs for 4 days and perform lightweight activity for 4 days. Patients will be observed for bleeding and significant abdominal pain postoperatively.

Justification of the clinical trial

EUS-LB has recently emerged as acceptable method to obtain liver tissue parenchyma for diagnostic purposes in both children and adult with abnormal liver chemistries. Several clinical studies have shown that obtaining liver tissue parenchyma by endoscopic ultrasonography is safe and reliable, compared to the traditional method, i.e. percutaneous approach.(2, 3, 5-14) In contrast to older methods (P-LB and TJ-LB), EUS-LB is targeted, with the ability to obtain liver tissue parenchyma from both hepatic lobes. In addition, EUS-LB can be combined with upper endoscopy as part of the evaluation for upper gastrointestinal symptoms/clinical presentation, and to evaluate for portal hypertension in cirrhotic patients. Moreover, a recent meta-analysis including 9 clinical studies reported an overall 93.6% histological diagnosis rate and a 2.3% adverse event rate with EUS-LB.(15) These studies, however, were flawed by their retrospective nature (only one study was prospective), variability in the demographics of patients undergoing EUS-LB, variability in the reported primary and secondary outcomes, variability in the reporting of insufficiency of specimens, variability in the core needle used, variability in the biopsy access route (trans-gastric vs. trans-duodenal), and variability in the biopsy site (right and left lobes vs. right lobe vs. left lobe). Our proposed clinical trial aims to examine the safety and efficacy of EUS-LB vs. P-LB in a prospective fashion under more stringent conditions. It is our hope that this prospective clinical trial will better define those who are ideal candidates for EUS-LB.

Study Statistics n. Primary outcome variable. o. Secondary outcome variables. p. Statistical plan including sample size justification and interim data analysis.

q. Early stopping rules.

1. Main outcomes measures are to assess EUS-LB vs. P-LB outcomes such as bleeding, pain, other complications after biopsies, tissue diagnosis.
2. Secondary outcome variable s will analyze demographic variables compared to outcomes and method
3. The investigators searched the literature and found only one prospective study comparing the safety and efficacy of EUS-LB vs. P-LB. In that study, it is unclear how the sample size was calculated. For the purposes of our proposed prospective clinical trial, our primary outcome measure is the number of complete portal tract(s) obtained per liver biopsy procedure. According to the most recent American Association for the Study of Liver Diseases (AASLD), an adequate liver biopsy for pathological interpretation is defined as a liver biopsy with ≥12 complete portal tracts. The investigators have designed a table showing variability of sample size calculations based on the assumed % of patients with ≥12 complete portal tracts in each group (i.e. EUS-LB vs. P-LB). For this study, the sample size is calculated based on the assumption that 90% of patients in the EUS-LB group will have liver biopsies with ≥12 complete portal tracts and 60% of patients in the P-LB will have liver biopsies with ≥12 complete portal tracts. Assuming a two-sided type I error of alpha (α)=0.05, at least 80% power, and a 1:1 ratio of EUS-LB vs. P-LB group, the estimated sample size for this study is 38 patients per group (total n= 76).

ELIGIBILITY:
Inclusion Criteria:

* all patients ≥ 18 years of age
* subjects undergoing a liver biopsy for focal/diffuse abnormalities of the liver
* parenchymal disease or chronically elevated liver function tests
* for assessing degree of fibrosis in chronic liver diseases
* or any indication deemed as necessary per the hepatologist/physician

Exclusion Criteria:

* Age <18
* Coagulopathy (INR of ≥1.5 and/or platelet count ≤ 50,000)
* Use of anticoagulants and/or blood thinners within 24 hours before the planned procedure
* Liver lesions such as hemangioma, echinococcal cyst or vascular tumors,
* Pregnancy,
* Uncooperative patients
* Any other condition or abnormalities that, in the opinion of the referring hepatologist or the advanced endoscopist, may compromise the safety of the patient or interfere with the patient participating in or completing the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
portal tracts obtained | 1 year
  the number of complete portal tract obtained in a biopsy between EUS vs. the percutaneous approach.

SECONDARY OUTCOMES:
Length of liver specimen. | 1 year
  the length will be measured in centimeters and the number of fragments noted
Pain score | Score will be calculated subjectively at the time of discharge after the biopsy and again in 24-48 hours after the procedure
  Pain scale used will be 1-10, 1 being no pain and 10 being the worst pain possible
Opiates consumed (in milligrams) per patients | This will be recorded at the time of discharge after the biopsy and again in 24-48 hours after the procedure
  Investigators will record how much and what kind of opiates the patient required to take after the procedure is complete. Investigators will also record the information of any additional opiates that the person required after the procedure in 24-48 hours duration
Readmission rate related to the procedure | Investigators will follow up the patient in 1 week duration to note any adverse events/complication that might have caused patient to get admitted to the hospital
  Here investigators will look for any events or complications after the procedure requiring admission to the hospital
Details of the liver biopsy procedure | Investigators will follow up and obtain this information within 1 month after the procedure
  Details such as the type of needle used during the procedure, amount of anesthesia required during the procedure and the total time spent during the procedure by the physician is recorded for comparison
Number of needle passes needed to obtain adequate sample. | Investigators will follow up and obtain this information within 1 month after the procedure
  For both percutaneous and EUS guided liver biopsies, investigators will calculate the number of passes that were necessary to obtain adequate sample by the surgeon which is available in the procedure note
Time for hospital stay per patient | Investigators will follow up and obtain this information within 1 month after the procedure
  Investigators will calculate the total time from the time of admission to the hospital to the discharge for each procedure performed to obtain the liver biopsy through chart review.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rockey DC, Caldwell SH, Goodman ZD, Nelson RC, Smith AD; American Association for the Study of Liver Diseases. Liver biopsy. Hepatology. 2009 Mar;49(3):1017-44. doi: 10.1002/hep.22742. No abstract available. PMID 19243014
- [Background] Diehl DL, Johal AS, Khara HS, Stavropoulos SN, Al-Haddad M, Ramesh J, Varadarajulu S, Aslanian H, Gordon SR, Shieh FK, Pineda-Bonilla JJ, Dunkelberger T, Gondim DD, Chen EZ. Endoscopic ultrasound-guided liver biopsy: a multicenter experience. Endosc Int Open. 2015 Jun;3(3):E210-5. doi: 10.1055/s-0034-1391412. Epub 2015 Feb 27. PMID 26171433
- [Background] Shah ND, Sasatomi E, Baron TH. Endoscopic Ultrasound-guided Parenchymal Liver Biopsy: Single Center Experience of a New Dedicated Core Needle. Clin Gastroenterol Hepatol. 2017 May;15(5):784-786. doi: 10.1016/j.cgh.2017.01.011. Epub 2017 Jan 23. No abstract available. PMID 28126424
- [Background] Nieto J, Khaleel H, Challita Y, Jimenez M, Baron TH, Walters L, Hathaway K, Patel K, Lankarani A, Herman M, Holloman D, Saab S. EUS-guided fine-needle core liver biopsy sampling using a novel 19-gauge needle with modified 1-pass, 1 actuation wet suction technique. Gastrointest Endosc. 2018 Feb;87(2):469-475. doi: 10.1016/j.gie.2017.05.013. Epub 2017 May 24. PMID 28551024
- [Background] Krupa L, Staron R, Pajak J, Lammert F, Krawczyk M, Gutkowski K. Secondary systemic amyloidosis diagnosed by endoscopic ultrasound-guided liver biopsy. J Gastrointestin Liver Dis. 2018 Mar;27(1):101-102. doi: 10.15403/jgld.2014.1121.271.kru. No abstract available. PMID 29557423
- [Background] Fally M, Nessar R, Behrendt N, Clementsen PF. Endoscopic Ultrasound-Guided Liver Biopsy in the Hands of a Chest Physician. Respiration. 2016;92(1):53-5. doi: 10.1159/000446924. Epub 2016 Jun 8. PMID 27287428
- [Background] Parekh PJ, Majithia R, Diehl DL, Baron TH. Endoscopic ultrasound-guided liver biopsy. Endosc Ultrasound. 2015 Apr-Jun;4(2):85-91. doi: 10.4103/2303-9027.156711. PMID 26020041
- [Background] Lee YN, Moon JH, Kim HK, Choi HJ, Choi MH, Kim DC, Lee TH, Lee TH, Cha SW, Kim SG, Kim YS. Usefulness of endoscopic ultrasound-guided sampling using core biopsy needle as a percutaneous biopsy rescue for diagnosis of solid liver mass: Combined histological-cytological analysis. J Gastroenterol Hepatol. 2015 Jul;30(7):1161-6. doi: 10.1111/jgh.12922. PMID 25684303
- [Background] Johal AS, Khara HS, Maksimak MG, Diehl DL. Endoscopic ultrasound-guided liver biopsy in pediatric patients. Endosc Ultrasound. 2014 Jul;3(3):191-4. doi: 10.4103/2303-9027.138794. PMID 25184126
- [Background] Nakai Y, Samarasena JB, Iwashita T, Park DH, Lee JG, Hu KQ, Chang KJ. Autoimmune hepatitis diagnosed by endoscopic ultrasound-guided liver biopsy using a new 19-gauge histology needle. Endoscopy. 2012;44 Suppl 2 UCTN:E67-8. doi: 10.1055/s-0031-1291567. Epub 2012 Mar 6. No abstract available. PMID 22396285
- [Background] Vegesna A, Nazir A, Chung CY, Kane S, Thomas R, Miller L. Acoustic liver biopsy in patients with hepatitis C and advanced liver fibrosis using endoscopic ultrasound. Dig Dis Sci. 2011 Oct;56(10):3053-7. doi: 10.1007/s10620-011-1670-6. Epub 2011 Apr 1. PMID 21455673
- [Background] Andanappa HK, Dai Q, Korimilli A, Panganamamula K, Friedenberg F, Miller L. Acoustic liver biopsy using endoscopic ultrasound. Dig Dis Sci. 2008 Apr;53(4):1078-83. doi: 10.1007/s10620-008-0211-4. Epub 2008 Feb 13. PMID 18270828
- [Background] Hollerbach S, Willert J, Topalidis T, Reiser M, Schmiegel W. Endoscopic ultrasound-guided fine-needle aspiration biopsy of liver lesions: histological and cytological assessment. Endoscopy. 2003 Sep;35(9):743-9. doi: 10.1055/s-2003-41593. PMID 12929021
- [Background] Mohan BP, Shakhatreh M, Garg R, Ponnada S, Adler DG. Efficacy and safety of EUS-guided liver biopsy: a systematic review and meta-analysis. Gastrointest Endosc. 2019 Feb;89(2):238-246.e3. doi: 10.1016/j.gie.2018.10.018. Epub 2018 Oct 31. PMID 30389469